CLINICAL TRIAL: NCT02496260
Title: Biomarkers and Cardiac MRI as Early Indicators of Cardiac Exposure
Brief Title: Biomarkers and Cardiac MRI as Early Indicators of Cardiac Exposure Following Breast Radiotherapy
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Dr. Eleanor Walker, Senior Staff Physician, Henry Ford Health System
Other Study IDs: 9481
Record Dates: First submitted 2015-06-23; First posted 2015-07-14 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Magnetic resonance imaging; Cardiac function; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of approximately 20 ml of blood will be performed by venipuncture at the specified time points. When possible, blood collection will be coordinated with other routine blood studies. These blood samples will be drawn at the clinical blood drawing station in the Radiation Oncology department.
  For fibrosis and left ventricular dysfunction, biomarkers include galectin-3 and NT-Pro brain natriuretic peptide. For myocyte destruction, troponin; for inflammation and oxidative stress, C-reactive protein, myeloperoxidase, and growth differentiation factor. Additional blood will be collected and stored for future assessment of other candidate biomarkers.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Research Cardiac MRI — Cardiac MRI has increased use in evaluating structural and functional cardiac pathologies. For detection of coronary artery disease, MRI outperforms SPECT and dobutamine stress echocardiography for the detection of ischemia. MRI also can detect wall-motion abnormalities and other dysfunction. Dynamic contrast-enhanced MRI (DCE-MRI) can evaluate microvascular parameters such as vessel permeability and fluid volume fraction as an assessment of tissue perfusion. Cardiac MRI holds promise for early detection of subclinical cardiac abnormalities after radiotherapy and could potentially identify patients for intervention to prevent cardiac events. All patients will follow the protocol calendar requiring research MRIs, but will receive standard radiation treatment determined by their physician. Treatment will not be altered based on MRI.
Procedure: Biomarkers — We have identified potential candidates based on other processes affecting heart function in a way similar to probable mechanisms of RT-related injury. For fibrosis and left ventricular dysfunction, these include galectin-3 and N-terminal-Pro brain natriuretic peptide. For myocyte destruction, troponin; for inflammation and oxidative stress, C-reactive protein, myeloperoxidase, and growth differentiation factor 15. Additional blood will be collected and stored for future assessment of other candidate biomarkers.
  All patients will follow the calendar of protocol required research blood draws for biomarker collection, but will receive standard radiation treatment as clinically indicated by their physician. Treatment will not be altered based upon the data collected from these samples.

SUMMARY:
Radiotherapy plays an integral role in breast cancer therapy. Multiple randomized studies have demonstrated decreased local-regional recurrence rates and decreased breast-cancer mortality. However, balanced with this survival benefit is the potential toxicity of the treatment itself. In particular, cardiac effects of radiotherapy have been a concern and an area of research for the past 20 years. From long-term follow up of patients with lymphoma, it is known that radiotherapy can lead to increased risk of myocardial infarction, valvular dysfunction, systolic and diastolic function abnormalities, and heart failure among cancer-survivors. Patients with breast cancer receive lower doses to smaller volumes of the heart, but they also have an excellent long-term survival, so it is crucial to study the effects of low dose radiotherapy. Indeed, a recent study suggests that these effects can be seen within the first 5 years after treatment, and that there is no dose threshold. This study aims to develop imaging and blood biomarkers of cardiac exposure, as a first step to identifying patients at increased risk for cardiac effects, so they can be targeted for close monitoring and early intervention, potentially with statins or ACE inhibitors. Additionally, by characterizing a time-course and radiation dose-volume relationship, potentially real-time modifications can be made to RT field design for patients sensitive to RT effects. Finally, this information can be incorporated into better designs of treatment plans for future patients.

DETAILED DESCRIPTION:
Radiotherapy plays an integral role in breast cancer therapy. Multiple randomized studies have demonstrated decreased local-regional recurrence rates and decreased breast-cancer mortality. However, balanced with this survival benefit is the potential toxicity of the treatment itself. In particular, cardiac effects of radiotherapy have been a concern and an area of research for the past 20 years. From long-term follow up of patients with lymphoma, it is known that radiotherapy can lead to increased risk of myocardial infarction, valvular dysfunction, systolic and diastolic function abnormalities, and heart failure among cancer-survivors. Patients with breast cancer receive lower doses to smaller volumes of the heart, but they also have an excellent long-term survival, so it is crucial to study the effects of low dose radiotherapy. Indeed, a recent study suggests that these effects can be seen within the first 5 years after treatment, and that there is no dose threshold. The investigators hypothesize that they can develop imaging and blood biomarkers of cardiac exposure, as a first step to identifying patients at increased risk for cardiac effects. These patients can then be targeted for close monitoring and early intervention, potentially with statins or ACE inhibitors. Additionally, by characterizing a time-course and radiation dose-volume relationship, potentially real-time modifications can be made to RT field design for patients sensitive to RT effects. Finally, this information can be incorporated into better designs of treatment plans for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive RT for left-sided breast cancer and can have a contrast-enhanced MRI are eligible.

Exclusion Criteria:

* Patients who have a contraindication to contrast-enhanced MRI are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pilot study of patients receiving radiotherapy for left-sided breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of patients in which cardiac MRI indicated subclinical cardiac abnormalities after radiotherapy that correlated with cardiac events | One year
  The study aims to characterize longitudinal changes in imaging characteristics of cardiac damage. Cardiac MRI endpoints will include myocardial edema, microvascular dysfunction, myocardial fibrosis, and subclinical impairment of systolic and diastolic function.

SECONDARY OUTCOMES:
Number patients in which blood and serum biomarkers were identified that correlated with cardiac damage due to radiation | One year
  The study aims to characterize longitudinal changes in potential early biomarkers of cardiac damage. Biomarker endpoints derived from blood or its components include measuring levels of galectin-3, NT-Pro brain natriuretic peptide, troponin, C-reactive protein, myeloperoxidase, and growth differentiation factor 15.
Number of unique biomarkers identified that were associated with radiation related cardiac injury | One year
  Biomarker endpoints derived from blood or its components include measuring levels of galectin-3, NT-Pro brain natriuretic peptide, troponin, C-reactive protein, myeloperoxidase, and growth differentiation factor 15. Additional biomarkers may be included as the research in those fields progresses during the conduct of this clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Morris ED, Ghanem AI, Pantelic MV, Walker EM, Han X, Glide-Hurst CK. Cardiac Substructure Segmentation and Dosimetry Using a Novel Hybrid Magnetic Resonance and Computed Tomography Cardiac Atlas. Int J Radiat Oncol Biol Phys. 2019 Mar 15;103(4):985-993. doi: 10.1016/j.ijrobp.2018.11.025. Epub 2018 Nov 22. PMID 30468849